CLINICAL TRIAL: NCT01996644
Title: A Double Blind Clinical Trial of DCS for Food Anxiety for Patients With Anorexia and Bulimia Nervosa
Brief Title: A Double Blind Clinical Trial of DCS for Food Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201212062; F31MH096433-01 (NIH)
Record Dates: First submitted 2013-11-18; First posted 2013-11-27 (Estimated); Results first posted 2018-03-27 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Anorexia and Bulimia Nervosa
Keywords: Anorexia, Bulimia, Anxiety, Exposure
MeSH Terms: conditions — Anorexia; Bulimia Nervosa; Bulimia; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Setraline (Experimental): 250 mg DCS (setraline) versus placebo plus exposure
  Interventions: Drug: Setraline
- placebo (Placebo Comparator): Placebo group plus exposure
  Interventions: Drug: Placebo vs Setraline

INTERVENTIONS:
Drug: Placebo vs Setraline — Placebo
  Other Names: Placebo
  Arms: placebo
Drug: Setraline — 250mg DCS
  Arms: Setraline

SUMMARY:
This is a pilot study investigating if cycloserine (DCS; a learning enhancement medication) augments exposure therapy for food anxiety in patients with anorexia and bulimia nervosa. The investigators expect that (a) exposure therapy will reduce anxiety (b) anxiety will be reduced more in the DCS relative to placebo condition (c) participants in the DCS condition will have a greater increase in Body Mass Index.

DETAILED DESCRIPTION:
This study investigated if DCS vs placebo augmented food exposure in individuals with eating disorders.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Anorexia Nervosa, Bulimia Nervosa, Eating Disorder Not Otherwise Specified

Exclusion Criteria:

* Pregnant or planning on becoming pregnant
* Psychotic or Manic

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University, St Louis, Missouri, United States

REFERENCES:
- [Derived] Levinson CA, Rodebaugh TL, Fewell L, Kass AE, Riley EN, Stark L, McCallum K, Lenze EJ. D-Cycloserine facilitation of exposure therapy improves weight regain in patients with anorexia nervosa: a pilot randomized controlled trial. J Clin Psychiatry. 2015 Jun;76(6):e787-93. doi: 10.4088/JCP.14m09299. PMID 26132687

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 47 participants were enrolled in the study, but only 36 were randomized and given any medication or placebo (i.e., participants completed the assessment portion of the study but did not move to the active experimental portion of the study).
Groups:
- Setraline: 250 mg DCS (setraline)
  Sertaline
- Placebo: Placebo group
Period: Overall Study
Arm/Group | Setraline | Placebo
Started | 20 | 16
Completed | 20 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Setraline: 250 mg DCS (setraline) versus placebo
  Sertaline
- Total: Total of all reporting groups
Arm/Group | Setraline | Placebo | Total
Number analyzed (Participants) | 20 | 16 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 2 | 5
  Between 18 and 65 years | 17 | 14 | 31
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 26.10 [15 to 49] | 24.63 [14 to 60] | 25.44 [14 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 16 | 35
  Male | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 16 | 36
BMI [Mean (Standard Deviation); unit: kg/m^2] | 20.10 (2.13) | 20.44 (1.91) | 20.25 (2.09)

OUTCOME MEASURES:

1. Primary Outcome: Anxiety as Measured by the Subjective Units of Distress (Ranging From 1 to 100).
Description: Anxiety will be measured at 4 sessions, twice a week for two weeks. Anxiety is combined in a repeated measures ANOVA to give total anxiety decreased across condition.
  Anxiety was measured using the Subjective Units of Distress (ranging from 1 to 100), where 1 is no anxiety and 100 is the most anxiety ever experienced.
Time Frame: Twice a week for two weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Setraline: 250 mg DCS (setraline) versus placebo
  Placebo vs Setraline: Placebo
Arm/Group | Setraline | Placebo
Number analyzed (Participants) | 20 | 16
Units on a scale | 52.395 (5.493) | 58.983 (6.141)

2. Primary Outcome: Body Mass Index
Description: BMI will be measured twice a week for two weeks and once before starting the trial. BMI is combined in a repeated measures ANOVA to give total BMI difference across condition.Difference in BMI from Time 1 to Time 4 was outcome.
Time Frame: twice a week for two weeks and at initial assessment
Measure: Mean (Standard Deviation); unit: kg/m^2
Groups:
- Placebo: Placebo group
  Sertaline
Arm/Group | Setraline | Placebo
Number analyzed (Participants) | 20 | 16
kg/m^2 | .385 (.3) | .095 (.3)
Statistical Analysis 1: Comparison: Setraline vs Placebo; Test type: Superiority or Other; p = .043, ANOVA

3. Other Pre Specified Outcome: Fear of Food Measure
Description: The Fear of Food Measure (FOFM) was designed to assess three cognitive behavioral components related to mealtime anxiety. All items are rated on a 1 to 7 Likert-type scale ranging from "not at all" to "very much so." Higher values indicate worse outcomes. The first subscale is the anxiety about eating subscale, which was designed to assess trait levels of fear and anxiety surrounding eating and food. This subscale will be measured once before and after the trial (twice in 2 weeks). Each item (8 items totaled, each scored 1-7; max possible score is 56; min possible score is 8) was added for each time point and time points were averaged together for all participants for both time points.
Time Frame: Twice during 2 weeks
Population: All combined represents the total number of participants (n=40); however 4 participants withdrew. Analysis utilized data for 36 participants who started in participant flow, thus (n=36).
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- All Combined: Setraline and Placebo groups
Arm/Group | Setraline | Placebo | All Combined
Number analyzed (Participants) | 20 | 16 | 36
Units on a scale | 19.55 (5.6) | 21.22 (5.8) | 20.01 (5.7)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 1 year.
Description: There were no adverse events recorded for any participants who started or finished the study.
Arm/Group | Setraline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/16
Other Adverse Events (participants affected / at risk) | 0/20 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No